CLINICAL TRIAL: NCT07198568
Title: Relationship Between Swallowing Dynamics and Suprahyoid Muscle Activity in Sarcopenic Dysphagia
Status: Recruiting | Type: Observational
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Joa KyungLim, M.D. PhD., Inha University Hospital
Other Study IDs: 2024-04-012
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Sarcopenia in Elderly; Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysphagic group: -Dysphagic group: Participants with a Penetration Aspiration score (PAS) of 3 points or higher that observed by Videofluoroscopic swallowing study were considered to have dysphagia
  Interventions: Diagnostic Test: Surface electromyography; Diagnostic Test: Videofluoroscopic swallowing study (VFSS)
- Non-dysphagic group: Participants with a Penetration Aspiration score (PAS) of 2 points or lower that observed by Videofluoroscopic swallowing study
  Interventions: Diagnostic Test: Surface electromyography; Diagnostic Test: Videofluoroscopic swallowing study (VFSS)

INTERVENTIONS:
Diagnostic Test: Surface electromyography — A previous other study has examined the suprahyoid muscle activity patterns in sarcopenic dysphagia patients using surface electromyography (sEMG). However, there was a lack of research analyzing the swallowing dynamics of sarcopenic dysphagia alongside Videofluoroscopic Swallowing Study (VFSS). VFSS enables the observation of swallowing in phases, offering a crucial method for assessing the presence of dysphagia and identifying the specific phases where dysphagia occurs. Therefore, the present study aims to investigate the characteristics of sarcopenic dysphagia across phases using sEMG and VFSS. Additionally, the investigators aim to analyze the relationship between suprahyoid muscle activity patterns and swallowing dynamics utilizing these modalities.
Diagnostic Test: Videofluoroscopic swallowing study (VFSS) — VFSS enables the observation of swallowing in phases, offering a crucial method for assessing the presence of dysphagia and identifying the specific phases where dysphagia occurs. The investigators will utilize Videofluoroscopic Dysphagia Scale (VDS), that composed of fourteen categories, which can be divided into oral and pharyngeal phases to assess scores based on VFSS results. The oral phase composed of 7 items (lip closure, bolus formation, mastication, apraxia, tongue-to-palate contact, premature bolus loss, and oral transit time). The pharyngeal phase also included 7 items (triggering of pharyngeal swallowing, vallecular residues, pyriform sinus residues, laryngeal elevation, coating of pharyngeal wall, pharyngeal transit time, and aspiration). VDS can assess the components of dysphagia in such detail. Therefore, investigators can evaluate the etiology of dysphagia more precisely.

SUMMARY:
Sarcopenic dysphagia is defined as swallowing difficulty among the elderly due to the loss of whole body skeletal and swallowing muscle mass and function. However, the pathophysiology and dynamics of swallowing in sarcopenic dysphagia have been poorly investigated. Therefore, the present study aims to investigate the characteristics of sarcopenic dysphagia using the Videofluoroscopic study (VFSS) focusing on each phase of dysphagia, and surface Electromyography (surface EMG) to assess suprahyoid muscle activity.

In sarcopenic dysphagia, impairments will occur in both the oral and pharyngeal phases, particularly affecting bolus formation, premature bolus spillage and laryngeal elevation during swallowing due to the loss of swallowing muscle mass and function. These changes will be considered to have led to an change of duration and amplitude of suprahyoid muscle activity measured via surface EMG.

DETAILED DESCRIPTION:
Measuring the muscle activity of the suprahyoid muscles presents a challenge due to their location, which is difficult to access. Despite this difficulty, surface Electromyography (sEMG) is an effective method for assessing the electrical activity of the suprahyoid muscles. sEMG is a non-invasive, portable, and cost-effective technique that records activity within the electrode detection area. It has been suggested as a diagnostic tool for identifying dysphagia. Several studies have demonstrated that specific patterns in the sEMG of suprahyoid muscles, including duration and amplitude, exhibit distinct characteristics attributable to various etiologies.

A previous study has examined the suprahyoid muscle activity patterns in sarcopenic dysphagia patients using sEMG. However, there was a lack of research analyzing the swallowing dynamics of sarcopenic dysphagia alongside Videofluoroscopic Swallowing Study (VFSS). VFSS enables the observation of swallowing in phases, offering a crucial method for assessing the presence of dysphagia and identifying the specific phases where dysphagia occurs.

Therefore, the present study aims to investigate the characteristics of sarcopenic dysphagia across phases using sEMG and VFSS. Additionally, Investigators aim to analyze the relationship between suprahyoid muscle activity patterns and swallowing dynamics utilizing these modalities.

Videofluoroscopic swallowing study (VFSS) will done for all participants to evaluate swallowing function. The VFSS procedure followed the Logemann protocol and will be supervised by a rehabilitation physician and an occupational therapist. Another physician will observe and score the test without having access to the patient's personal details.

During the VFSS, participants will seat upright in a chair, swallowing images of the lateral projection will be obtained from participants. The participants undergo swallowing trials with varying viscosities, including semiliquid, semisolid, solid, and thin liquids (2cc, 5cc, 10cc). All trials are mixed with an undiluted liquid barium solution, barium sulfate. During the procedure, participants will undergo progressively thicker food, starting from liquids and advancing to solid materials. Following the protocol, liquid 2 cubic centimeter (cc) trial will precede to the 5cc trial. If, the 2cc trial indicated aspiration and the physician determined there was a high risk for aspiration, next step of trial can be skipped and the VFSS will be stopped. If, a large amount of aspiration occurred, the VFSS will be halted, and the participant will encouraged to expectorate the food material.

The activity of suprahyoid muscles will be recorded using a surface electromyography. Pairs of disposable self-adhesive electrodes will fixed to the skin surface of the suprahyoid muscles. The electrodes positioned symmetrically between the hyoid bone and the chin, with a center-to-center distance of 20mm. Before attaching, participants will seated upright in a chair and the skin surface will be cleaned using alcohol swabs. After attaching the electrodes, participant instructed to open their jaw as wide as they could for 10 seconds to measure the amplitude, which can be used as a reference for normalization. The amplitude of sEMG is influenced by various tissue conditions. Therefore, normalization based on a reference muscle contraction is necessary to compare amplitudes between individuals. Subsequently, participants will received 2ml of water on the floor of the mouth using a syringe, and will be instructed to swallow under the guidance of a rehabilitation physician. Each participant undergo three trials of water swallowing, separated by 30 seconds intervals.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older who underwent VFSS to evaluate the presence of dysphagia
* Patient who diagnosed with sarcopenia based on the cutoff values of the Asian Working Group for Sarcopenia (AWGS) 2019
* Cognitive ability to follow instructions for Videofluoroscopic swallowing study, surface electromyography.

Exclusion Criteria:

* History of cerebral hemorrhage or cerebral infarction
* History of neuromuscular diseases that could lead to dysphagia such as Parkinson's disease, amyotrophic lateral sclerosis, Guillain-Barre disease
* History of Tracheostomy
* History of oropharyngeal cancer
* History of esophageal structural disease that could lead to dysphagia
* History of connective tissue disease
* History of cervical surgical procedure
* Cognitive impairment who cannot follow instructions for Videofluoroscopic swallowing study, surface electromyography

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted at an Inha University Hospital, tertial general hospital in Republic of Korea and referred to the department of physical and rehabilitation medicine to evaluate for presence of dysphagia and meet the inclusion criteria specified above.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Amplitude of suprahyoid muscle activity: Surface electromyography data | Baseline
  The measurement parameters included the mean and maximum amplitudes of suprahyoid muscle activation during swallowing. Amplitude values were normalized relative to the amplitude observed during jaw opening contraction (JOC). Both mean and maximum amplitudes were subsequently expressed as percentages of the jaw opening contraction (%JOC).
Total duration of suprahyoid muscle activity: Surface electromyography data | Baseline
  The onset of swallowing was defined as the point at which a distinct visual increase in sEMG activity above the background level was observed and the end point of swallowing was determined as the moment when the sEMG trace returned to within +2 standard deviations (SDs) of the baseline amplitude level. The baseline amplitude was calculated as the average amplitude during a 1 second period at rest from the start of the sEMG trace.
Onset to peak duration of suprahyoid muscle activity: Surface electromyography data | Baseline
  duration from the swallowing onset to the maximum amplitude point
Peak to onset duration of suprahyoid muscle activity: Surface electromyography data | Baseline
  duration from the maximum amplitude point to the end of the swallowing

SECONDARY OUTCOMES:
Videofluoroscopic dysphagia scale (VDS) that assessed by Videofluoroscopic swallowing study (VFSS) | baseline
  VDS is composed of fourteen categories, which can be divided into oral and pharyngeal phases to assess scores based on VFSS results. The oral phase composed of 7 items (lip closure, bolus formation, mastication, apraxia, tongue-to-palate contact, premature bolus loss, and oral transit time). The pharyngeal phase also included 7 items (triggering of pharyngeal swallowing, vallecular residues, pyriform sinus residues, laryngeal elevation, coating of pharyngeal wall, pharyngeal transit time, and aspiration). The scoring system of VDS ranges from 0 to 100, with up to 40 points for oral phase, and 60 points for pharyngeal phase. Higher scores correspond to more severe dysphagia.
Penetration aspiration scale (PAS) that assessed by Videofluoroscopic swallowing study (VFSS) | Baseline
  The Penetration-Aspiration Scale (PAS), which consists of 8 points, is used to measure the severity of airway invasion events and the patient's responses during VFSS. The scoring system of PAS ranges from 1 to 8. Higher scores correspond to more severe dysphagia.
Parramatta Hospital's assessment of dysphagia that assessed by Videofluoroscopic swallowing study (VFSS) | Baseline
  The Parramatta Hospitals Assessment of Dysphagia provides a quantitative rating of swallowing. It is composed of fourteen aspects of bulbar and swallowing function (the level of alertness, respiratory function, comprehension, expression, lip, tongue, palatal motor function, gag reflex, phonation, cough, preparatory, oral and pharyngeal stages of swallowing, and tolerance for differing food consistencies). The scoring system of Parramatta Hospital's assessment of dysphagia ranges from 20 to 100. Lower scores correspond to more severe dysphagia
American Speech-Language-Hearing Association National Outcome Measurement System swallowing scale (ASHA NOMS scale) that assessed by Videofluoroscopic swallowing study (VFSS) | Baseline
  The ASHA-NOMS scale assesses the functional level of swallowing. This measurement indicates the level of supervision necessary for feeding and suggests the appropriate diet type, with scores from 1 to 7. Lower scores correspond to more severe dysphagia.

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, Jung-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sakai K, Nakayama E, Rogus-Pulia N, Takehisa T, Takehisa Y, Urayama KY, Takahashi O. Submental Muscle Activity and Its Role in Diagnosing Sarcopenic Dysphagia. Clin Interv Aging. 2020 Oct 21;15:1991-1999. doi: 10.2147/CIA.S278793. eCollection 2020. PMID 33116453
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Wakabayashi H, Sashika H, Matsushima M. Head lifting strength is associated with dysphagia and malnutrition in frail older adults. Geriatr Gerontol Int. 2015 Apr;15(4):410-6. doi: 10.1111/ggi.12283. Epub 2014 Apr 1. PMID 24690326
- [Background] Shapiro J. Evaluation and treatment of swallowing disorders. Compr Ther. 2000 Fall;26(3):203-9. doi: 10.1007/s12019-000-0010-0. PMID 10984826
- [Background] Vaiman M, Eviatar E. Surface electromyography as a screening method for evaluation of dysphagia and odynophagia. Head Face Med. 2009 Feb 20;5:9. doi: 10.1186/1746-160X-5-9. PMID 19232090
- [Background] Monaco A, Cattaneo R, Spadaro A, Giannoni M. Surface electromyography pattern of human swallowing. BMC Oral Health. 2008 Mar 26;8:6. doi: 10.1186/1472-6831-8-6. PMID 18366770
- [Background] Shaw SM, Martino R. The normal swallow: muscular and neurophysiological control. Otolaryngol Clin North Am. 2013 Dec;46(6):937-56. doi: 10.1016/j.otc.2013.09.006. Epub 2013 Oct 23. PMID 24262952
- [Background] Tamura F, Kikutani T, Tohara T, Yoshida M, Yaegaki K. Tongue thickness relates to nutritional status in the elderly. Dysphagia. 2012 Dec;27(4):556-61. doi: 10.1007/s00455-012-9407-z. Epub 2012 Apr 27. PMID 22538556
- [Background] Dellis S, Papadopoulou S, Krikonis K, Zigras F. Sarcopenic Dysphagia. A Narrative Review. J Frailty Sarcopenia Falls. 2018 Mar 1;3(1):1-7. doi: 10.22540/JFSF-03-001. eCollection 2018 Mar. PMID 32300688
- [Background] Yoshimura N, Muraki S, Oka H, Iidaka T, Kodama R, Kawaguchi H, Nakamura K, Tanaka S, Akune T. Is osteoporosis a predictor for future sarcopenia or vice versa? Four-year observations between the second and third ROAD study surveys. Osteoporos Int. 2017 Jan;28(1):189-199. doi: 10.1007/s00198-016-3823-0. Epub 2016 Nov 24. PMID 27885410
- [Background] Woo J, Leung J, Morley JE. Defining sarcopenia in terms of incident adverse outcomes. J Am Med Dir Assoc. 2015 Mar;16(3):247-52. doi: 10.1016/j.jamda.2014.11.013. Epub 2014 Dec 23. PMID 25548028
- [Background] Palmer K, Onder G, Cesari M. The geriatric condition of frailty. Eur J Intern Med. 2018 Oct;56:1-2. doi: 10.1016/j.ejim.2018.09.011. Epub 2018 Sep 22. No abstract available. PMID 30253892
- [Background] de Sire A, Giachero A, DE Santi S, Inglese K, Solaro C. Screening dysphagia risk in 534 older patients undergoing rehabilitation after total joint replacement: a cross-sectional study. Eur J Phys Rehabil Med. 2021 Feb;57(1):131-136. doi: 10.23736/S1973-9087.20.06321-2. Epub 2020 Jun 26. PMID 32594668
- [Background] Abdullah B, Wolbring G. Analysis of newspaper coverage of active aging through the lens of the 2002 World Health Organization Active Ageing Report: A Policy Framework and the 2010 Toronto Charter for Physical Activity: A Global Call for Action. Int J Environ Res Public Health. 2013 Dec 5;10(12):6799-819. doi: 10.3390/ijerph10126799. PMID 24317386